CLINICAL TRIAL: NCT05092074
Title: Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) for Patients With Hepatitis C Virus Infection: Real-world Effectiveness and Safety in Taiwan
Brief Title: Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) for Patients With Hepatitis C Virus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202109016RIND
Record Dates: First submitted 2021-10-03; First posted 2021-10-25 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C Virus Infection; Treatment Side Effects; Adherence, Treatment; Effect of Drug
Keywords: Hepatitis C virus; Sofosbuvir; Velpatasvir; Voxilaprevir
MeSH Terms: conditions — Hepatitis C; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. 5 mL of whole blood to detect the HCV viral resistance profiles (NS3 and NS5A regions) in all participants before SOF/VEL/VOX treatment
  2. 5 mL of whole blood to detect the HCV viral resistance profiles (NS3 and NS5A regions) in participants who fail to respond to SOF/VEL/VOX treatment after off-therapy 12 weeks of observation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vosevi 400/100/100 Oral Tablet — Sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX, Vosevi) 400/100/100 oral tablet: 1 table per os per day for 12 weeks

SUMMARY:
The investigators aim to assess the effectiveness and safety of sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) for 12 weeks in hepatitis C virus (HCV)-infected patients who fail to prior NS5A-containing DAA regimens and HCV genotype 1a and 3 patients who fail to prior non-NS5A-containing DAA regimen in Taiwan on a basis of a multicenter observational study.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a global health problem and it is estimated that about 71 million people are HCV carriers worldwide. Based one the excellent efficacy and safety, interferon (IFN)-free direct-acting antiviral agents (DAAs) have become the standard of care (SOC) for the care of HCV. Currently, about 10 different DAA regimens have been approved by FDA and EMA for the treatment of HCV, the sustained virologic response (SVR) rates are generally more than 95% by these treatment.

Despite the efficacy and safety are excellent in patients receiving DAAs for HCV, about 1%-5% of these patients fail to successfully clear virus by DAA treatment. Retreating patients who fail to respond to DAAs with more potent DAAs would be of paramount importance for treating physicians and patients. Even since 2017, an estimated of 110,000 to 120,000 viremic patients in Taiwan have received governmental reimbursement with DAA treatment. Based on a recent report from National Hepatitis C Program (NHCP) office, about 2% of subjects in Taiwan have virologic failures to DAA treatment, which implies that about 2,200 to 2,400 HCV-infected patients remain viremic with the currently approved first-line DAA therapies. Furthermore, the majority of them have been treated with HCV non-structural 5A (NS5A)-based DAA regimens. Sofosbuvir/velpatasvir/voxilaprevir, a pangenotypic DAA regimen, serves as a rescue therapy for HCV patients who do not respond to first-line DAA treatment. The phase 3 POLARIS-1 trial which retreated HCV patients who failed to respond to NS5A-containing DAAs with SOF/VEL/VOX for 12 weeks revealed that the SVR12 rate was 96%. Among patients without cirrhosis and with compensated cirrhosis, the SVR12 rates were 99% and 93%, respectively. In addition, the phase 3 POLARIS-4 trial which retreated HCV genotype 1a and 3 patients who failed to respond to non-NS5A-containing DAAs with SOF/VEL/VOC for 12 weeks in HCV revealed that the SVR12 rates were 98% and 94%, respectively. Because all patients enrolled in the POLARIS-1 and POLARIS-4 trials who failed to prior genotype-specific DAA regimens, data regarding the effectiveness and safety of SOF/VEL/VOX for patients who failed to prior pangenotypic DAA regimens remain elusive. Two small-scale real-world studies assessing the performance of SOF/VEL/VOX for 12 weeks in patients who failed to pangenotypic SOF/VEL or glecaprevir/pibrentasvir (GLE/PIB) revealed that SVR12 rates were 100% and 94%. Nonetheless, two real-world studies in Western countries showed that the SVR12 rates of SOF/VEL/VOX for 12 weeks ranged from 95%-96% for HCV patients who failed to prior DAA therapies.

Based on the approval of governmental reimbursement of SOF/VEL/VOX retreatment for HCV genotype 1-6 patients who fail to prior NS5A-containing DAA regimens and HCV genotype 1a and 3 patients who fail to prior non-NS5A-containing DAA regimen on September 1, 2021 in Taiwan, the investigators aim to conduct a multicenter observational study to assess the real-world effectiveness and safety of SOF/VEL/VOX for 12 weeks in these patients to provide a powerful evidence to optimize the clinical practice in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV) infection, defined as the presence of HCV RNA for ≥ 6 months
* Age ≥ 20 years
* Patients with any HCV genotype (genotype 1-6 or indeterminate genotype) who failed to NS5A-containing DAA regimen or patients with HCV genotype 1a or 3 who failed to non-NS5A-containing DAA regimen

Exclusion Criteria:

* Decompensated cirrhosis
* Patients who receive concomitant medications which are contraindicated for SOF/VEL/VOX, and who decline to stop or switch contraindicated concomitant medications
* Patients who receive therapeutic vaccination or other investigational agents for HCV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C virus-infected patients who are aged 20 years or more and who are not responded to a prior course of NA5A-containing DAA regimen (all viral genotypes) or to a prior course of non-NS5A-containing DAA regimen (viral genotype 1a or 3). Patients should have compensated liver diseases, and should not take co-medications which are contraindicated for use in the presence of SOF/VEL/VOX.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | A total of 24 weeks after the initiation of treatment (drug treatment for 12 weeks and off-treatment follow-up for additional 12 weeks)
  Number and percentage of participants who have undetectable serum level of HCV RNA at off-treatment week 12

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Director — National Taiwan University Hospital
Locations (15):
- Taiwan (15):
  - China Medical University Beigang Hospital, Beigang
  - Changhua Christian Hospital, Changhua
  - Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City
  - St. Martin De Porres Hospital, Chiayi City
  - Yang Ming Hospital, Chiayi City
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Dalin
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Chi-Mei Medical Center, Liouying, Liuying
  - Fu Jen Catholic University Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No